CLINICAL TRIAL: NCT03983005
Title: Observational, Prospective, Multicenter Study on the Diagnostic Accuracy, Safety and Tolerability, Predictors of Success of EUS-B-FNA in the Diagnosis of Malignant Parenchymal Lung Lesions
Brief Title: EUS-B-FNA in the Diagnosis of Malignant Parenchymal Lung Lesions
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Michele Mondoni, MD, Principal Investigator, University of Milan
Other Study IDs: EUS-B
Record Dates: First submitted 2019-06-01; First posted 2019-06-12 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Endoscopic ultrasound; EUS-B-FNA; Molecular analysis; Rapid on-site evaluation
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Needle aspirations
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with suspected lung cancer: Patients with pulmonary parenchymal lesions suspected for malignancy in contact or adjacent to the esophagus which can be sampled by EUS-B-FNA
  Interventions: Procedure: EUS-B-FNA

INTERVENTIONS:
Procedure: EUS-B-FNA — Endoscopic ultrasound with bronchoscope fine needle aspiration (EUS-B-FNA) is an endoscopic technique based on a trans-esophageal needle aspiration performed by an interventional pulmonologist with the echo-bronchoscope
  Other Names: Endoscopic ultrasound with bronchoscope fine needle aspiration

SUMMARY:
The aim of this study is to evaluate the diagnostic accuracy, safety and tolerability, predictors of success of EUS-B-FNA in the diagnosis of malignant parenchymal lung lesions.

The Investigators will also evaluated the adequacy of samples obtained for molecular analysis in patients with Non-Small Cell Lung Cancer (NSCLC)

DETAILED DESCRIPTION:
Lung cancer is by far the leading cause of cancer death among both men and women worldwide. Non-Small Cell Lung Cancer (NSCLC) represents about 80-90% of all lung cancers. Endoscopic ultrasound with bronchoscope fine needle aspiration (EUS-B-FNA) is a safe and accurate technique that has been mostly described for the diagnosis and the mediastinal nodal staging of NSCLC, as a complementary technique to endobronchial ultrasound trans-bronchial needle aspiration (EBUS-TBNA) or when EBUS-TBNA may be difficult and/or contraindicated for clinical reasons (e.g. excessive cough, respiratory failure etc).

Few retrospective studies evaluated the sensitivity and the safety of this technique in the diagnosis of parenchymal pulmonary lesions suspected for lung cancer, in contact or adjacent to the esophagus. Few data are available on the adequacy of the samples obtained by EUS-B-FNA for molecular analysis in NSCLC. The main predictors of success are still unclear.

The primary aim of this prospective study is to evaluate the diagnostic accuracy of EUS-B-FNA in the diagnosis of malignant parenchymal lung lesions. The Investigators will also evaluate the safety and tolerability of the technique, the main predictors of success and the adequacy of samples obtained for molecular analysis in patients with NSCLC

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a lung parenchymal lesion suspected for malignancy, in contact or adjacent to the esophagus at the CT scan (with or without mediastinal lymph adenopathies), requiring a pathological diagnosis:

  * which can not be sample by bronchoscopy/EBUS-TBNA or
  * with a previous not diagnostic bronchoscopy/EBUS-TBNA or
  * with clinical/anesthesiological contraindications to bronchoscopy/EBUS-TBNA or
  * with a previous nodal EUS-B-FNA not diagnostic/not adequate at the ROSE
* Patients with lung parenchymal lesions who are able to sign the informed consent for the study participation

Exclusion Criteria:

* Patients with lung parenchymal lesions of known etiology;
* Patients with lung parenchymal lesions in whom bronchoscopic ultrasound-guided trans- esophageal needle aspiration is contraindicated;
* Patients with lung parenchymal lesions who refuse/are not able to sign the informed consent for the study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a parenchymal lung lesion suspected for malignancy in contact or adjacent to the esophagus at the CT scan, who need a pathological diagnosis.
Sampling Method: Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of EUS-B-FNA in the detection of malignant pulmonary lesions | At study completion (expected February 2021)
  Diagnostic accuracy (i.e., sensitivity and specificity) of EUS-B-FNA in the diagnosis of malignant pulmonary parenchymal lesions, discriminating those with a malignant disease in comparison with those without the malignant disease. A specific unit of measure is not included, being the computation of the present outcome based on the absolute number of malignant/non malignant cases to the total number of diagnosed individuals.

SECONDARY OUTCOMES:
Absolute and relative frequency of adequate samples for molecular analysis in NSCLC following assessment by pathologist/molecular biologist | At study completion (expected February 2021)
  Proportional number (percentage) of samples obtained with EUS-B-FNA containing sufficient material (i.e. malignant cells) for molecular analysis in NSCLC following assessment by a pathologist/molecular biologist. A specific unit of measure is not included, being the computation of the present outcome based on the absolute number of malignant cells in the single sample.
Detection of predictors of successful aspirate based on the implementation of regression models | At study completion (expected February 2021)
  Implementation of regression models (logistic regression analysis) to detect variables related to a successful aspirate: anatomical (i.e. lung, lobe of the lesion), endoscopic (type of endoscope, type of needle, number of needle passes, needle aspiration technique), pathological (presence/absence of rapid on-site evaluation (ROSE), health personnel performing ROSE (i.e pathologist, respiratory physician, cytotechnician), pathological technique used for diagnosis and molecular analysis (smear, cell-block, liquid based cytology). A specific unit of measure is not included, being the computation of the present variables based on the measurement of absolute numbers not recorded with a specific unit of measure. The unit of measure is basically identified by the single element of the variable.
Safety (number of adverse events) of EUS-B-FNA through CTCAE v4.0 | Until 24 hours after the procedure
  Incidence rate and qualitative and quantitative description of adverse events in patients undergoing EUS-B-FNA. A specific unit of measure is not included, being the computation of the present outcome based on the absolute number of the adverse events detected by the attending physician.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Mondoni, MD, Principal Investigator — Respiratory Unit, ASST Santi Paolo e Carlo, San Paolo Hospital
Locations (4):
- Italy (4):
  - UO Pneumologia dell'Ospedale dell'Angelo, Mestre, Venice
  - Pulmonology Unit, AOU "Ospedali Riuniti"; Department of Biomedical Sciences and Public Health, Università Politecnica delle Marche, Ancona
  - Respiratory Unit, ASST Santi Paolo e Carlo, San Paolo Hospital, Department of Health Sciences, Università degli Studi di Milano, Milan
  - Unità Operativa Complessa di Pneumologia, Fondazione Policlinico Universitario A. Gemelli IRCCS, Università Cattolica del Sacro Cuore, Rome